CLINICAL TRIAL: NCT00797758
Title: Assessment of Reduction of Cord Blood Transplantation Toxicity by Using Reduced Intensity Conditioning in Patients With Acute Myeloid Leukemia.
Brief Title: Reduction of Cord Blood Transplantation Toxicity in Patients With Acute Myeloid Leukemia
Acronym: MINICORD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 060206
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Cord blood transplantation; Conditioning regimen; Acute myeloid leukaemia; SORROR comorbidity index; Quality of life; Innate immunity; Immune reconstitution post transplant; Umbilical Cord Blood Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Umbilical cord blood transplantation after reduced intensity conditioning
  Interventions: Other: Cord blood transplantation

INTERVENTIONS:
Other: Cord blood transplantation — Umbilical cord blood transplantation after reduced intensity conditioning

SUMMARY:
Multicentric evaluation of the reduction of unrelated cord blood transplantation (UCBT) toxicity by using reduced intensity conditioning (RIC) in patients with acute myeloid leukaemia.UCBT related mortality and morbidity were limiting factors for the development of this procedure in adults. Non myeloablative conditioning regimen showed promising results and prospective evaluation has to be developed to confirm these retrospective data.

DETAILED DESCRIPTION:
Individual meta-analysis is planned to compare geno-identical transplantation with myeloid-ablative or non myeloid-ablative conditioning with UCBT after RIC.

ELIGIBILITY:
Inclusion Criteria:

* Ages : 4 to 65
* De novo or secondary AML requiring allogeneic transplant
* No donor (related or unrelated) compatible 10/10
* Complete remission excepted CR1 with t(8;21) or inv (16) or t (15;17)
* Smouldering AML without progression
* Signed assent of recipient

Exclusion Criteria:

* If CR1: AML with with t(8;21) or inv (16) or t (15;17)
* Karnofsky < 50% - Clearance of creatinin < 40 ml/min
* Transaminases > 8 N
* Previous autologous or allogeneic transplantation within 6 month prior to the study (except if tandem)
* total body irradiation contra-indicating 2 Gy TBI
* local irradiation contra-indicating 2 Gy TBI

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Transplant related mortality | At 2 years

SECONDARY OUTCOMES:
Clinical efficiency (overall survival, event free survival, relapse incidence, acute and chronic GVHD incidence, graft failure, venoocclusive disease, interstitial pneumonia, infections, comorbidity score, quality of life and medico-economic impact) | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard RIO, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Département d'Hématologie et d'Oncologie Médicale, Hôtel-Dieu, Paris, France

REFERENCES:
- [Derived] Rio B, Chevret S, Vigouroux S, Chevallier P, Furst S, Sirvent A, Bay JO, Socie G, Ceballos P, Huynh A, Cornillon J, Francoise S, Legrand F, Yakoub-Agha I, Michel G, Maillard N, Margueritte G, Maury S, Uzunov M, Bulabois CE, Michallet M, Clement L, Dauriac C, Bilger K, Gluckman E, Ruggeri A, Buzyn A, Nguyen S, Simon T, Milpied N, Rocha V; Societe Francaise de Greffe de Moelle et de Therapie Cellulaire and Eurocord. Decreased nonrelapse mortality after unrelated cord blood transplantation for acute myeloid leukemia using reduced-intensity conditioning: a prospective phase II multicenter trial. Biol Blood Marrow Transplant. 2015 Mar;21(3):445-53. doi: 10.1016/j.bbmt.2014.11.009. Epub 2014 Nov 18. PMID 25460357